CLINICAL TRIAL: NCT04936711
Title: Randomized Prospective Interventional Study: Pain Relief After Laparoscopic Primary Hiatal Hernia Repair
Brief Title: Pain Relief After Hiatal Hernia Repair Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norton Thoracic Institute (Other)
Responsible Party: Principal Investigator, Leslie Munson, Research Program Manager, Norton Thoracic Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHX-21-500-157-50-18
Record Dates: First submitted 2021-05-19; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Shoulder Pain; Hiatal Hernia
Keywords: Shoulder pain; Hernia; Hernia surgery; Hernia repair; Hiatal hernia; Hiatal hernia surgery; Hiatal hernia repair; Post surgery pain
MeSH Terms: conditions — Shoulder Pain; Hernia, Hiatal; Hernia | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Back Massager Device + Standard Pain Treatment (Experimental): Resteck Shiatsu Neck and Back Massager (brand name), with recommended use for at least every 2 hours for at least 15 minutes on the first post-operative day and then every 4 hours for 2 days and then as needed.
  Standard pain treatment:
  1. Local anesthetic agent at the incision sites include: 0.5% Marcaine (10 cc) + 0.5% lidocaine and epinephrine (10 cc) (total volume: 20 cc)
  2. Morphine 2 mg: Intravenous administration every 2 hours or as needed, if unable to take pills by mouth
  3. Oxycodone 5 - 10 mg elixir: oral administration every 6 hours or as needed
  4. Tylenol 650 mg Tab: oral administration every 6 hours
  Interventions: Device: Resteck Shiatsu Neck and Back Massager
- Marcaine spray + Standard Pain Treatment (Active Comparator): 30cc of 0.25% Marcaine spray on the diaphragm at the end of surgery.
  Standard pain treatment:
  1. Local anesthetic agent at the incision sites include: 0.5% Marcaine (10 cc) + 0.5% lidocaine and epinephrine (10 cc) (total volume: 20 cc)
  2. Morphine 2 mg: Intravenous administration every 2 hours or as needed, if unable to take pills by mouth
  3. Oxycodone 5 - 10 mg elixir: oral administration every 6 hours or as needed
  4. Tylenol 650 mg Tab: oral administration every 6 hours
  Interventions: Drug: Marcaine
- Standard Pain Treatment (No Intervention): will receive standard pain treatment include local anesthetic agent at the incision sites + oral Tylenol and oral or IV opioid as breakthrough pain treatment postoperatively as needed.
  Standard pain treatment:
  1. Local anesthetic agent at the incision sites include: 0.5% Marcaine (10 cc) + 0.5% lidocaine and epinephrine (10 cc) (total volume: 20 cc)
  2. Morphine 2 mg: Intravenous administration every 2 hours or as needed, if unable to take pills by mouth
  3. Oxycodone 5 - 10 mg elixir: oral administration every 6 hours or as needed
  4. Tylenol 650 mg Tab: oral administration every 6 hours

INTERVENTIONS:
Device: Resteck Shiatsu Neck and Back Massager — back massager device sold on the market that can readily be purchased online or in store
  Arms: Back Massager Device + Standard Pain Treatment
Drug: Marcaine — Marcaine spray at incision site after closure
  Other Names: bupivacaine hydrochloride
  Arms: Marcaine spray + Standard Pain Treatment

SUMMARY:
Referred shoulder pain (pain felt when the problem is actually in a different location) is very common after laparoscopic (small, narrow cut) hernia surgery. The purpose of this study is to look at the effect of a simple back massager, which can be readily purchased online or in a store, in addition to the use of standard pain medications.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for primary hiatal hernia repair
* Adult 18 years of age or older
* Undergoing minimally invasive surgical technique

Exclusion Criteria:

* Recurrent hiatal hernia
* Children under the age of 18 years
* Undergoing open or hybrid surgical technique
* History of psychiatric disorder or chronic pain
* Has a post-operative complication (Grade > I on Calvien Dindo classification)
* Allergy to standard pain medication regimen (local anesthetics Marcaine, lidocaine, and epinephrine; morphine; oxycodone; Tylenol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score Pain Questionnaire | 2 years
  Pain score questionnaire to rate pain on a scale of 0 - 10, with 0 being no pain and 10 being the worst possible pain imaginable. The higher the score, the worse the outcome.
Opioid and Non-Opioid Usage Postoperative Period | 2 years
  Subject diary to list any medications taken for pain relief after surgery, and will list the following: name of medication, dose of medication, date and time medication taken

CONTACTS AND LOCATIONS:
Overall Officials: Sumeet K Mittal, MD, Principal Investigator — St. Joseph's Hospital and Medical Center, Norton Thoracic Institute
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mittal SK, Latorre-Rodriguez AR, Bremner RM. Shoulder pain after laparoscopic antireflux surgery: a single-center, randomized, open-label trial. Surg Endosc. 2025 Aug;39(8):5355-5366. doi: 10.1007/s00464-025-11939-3. Epub 2025 Jul 2. PMID 40603619